CLINICAL TRIAL: NCT03045575
Title: Objective Assessment of Physical Activity During Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 157512; 15-17054 (Other: University of California, San Francisco)
Record Dates: First submitted 2017-01-27; First posted 2017-02-07 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study designed to determine the feasibility and acceptability of objectively measuring physical activity, sedentary time, and sleep using the Fitbit Charge HR wristband. 50 patients who have been diagnosed with breast cancer and are planning to initiate chemotherapy will be invited to participate in this study, and we will measure general and breast-specific quality-of-life using Patient-Reported Outcomes Measurement Information System (PROMIS) measures for 3-6 months after completion of chemotherapy.

DETAILED DESCRIPTION:
Over 3.1 million women are currently living with a diagnosis of breast cancer in the United States (US), representing 41% of all female cancer survivors in the US. The increased breast cancer survival rate has necessitated a shift in cancer care toward developing interventions to empower patients to improve their quality-of-life, and perhaps prognosis, during and after treatment. Among women diagnosed with early-stage (I or II) breast cancer, around 40% will receive chemotherapy. Among women diagnosed with late-stage (III or IV), around 75% will receive chemotherapy. Adjuvant chemotherapy is associated with many side effects, including fatigue, nausea, disturbed sleep, decreased activity, and weight gain. Women receiving chemotherapy gain an average of 2.5 to 6.2 kg during therapy. Weight gain increases the risk of breast cancer recurrence and mortality, as well as cardiovascular disease, diabetes, and second primary cancers. Physical activity alleviates or reduces both short and long term treatment side effects of chemotherapy, including weight gain, and restores physical functioning in breast cancer patients. Additionally, randomized controlled trials in breast cancer patients have shown that adding exercise to chemotherapy programs can improve breast cancer outcomes.

Although there are many benefits of engaging in physical activity during cancer treatments, activity levels typically decline throughout treatment. Existing research has relied on self-reported activity levels, which is a poor measure of low-intensity activities and can only capture a periodic snap shot of activity levels. This study will provide objective physical activity data across the entirety of the patient's chemotherapy treatments. This in depth data will provide a new perspective on the patterns of activity levels and help to identify if there are critical times in which to intervene to prevent physical activity declines.

ELIGIBILITY:
Inclusion Criteria:

* have been diagnosed with breast cancer
* be planning to initiate chemotherapy for breast cancer at University of California, San Francisco (UCSF)
* be able to speak and read English, or have a family member or friend who can assist in translating and completing surveys in English
* be able to walk unassisted
* be able to navigate websites, fill out forms on the web, communicate by email, and have regular access to the internet

Exclusion Criteria:

* We will exclude individuals who cannot speak or read English unless they have a friend or family member who can assist in translating and completing quality of life surveys in English. In addition, the Fitbit® requires the ability to connect to the Internet and input data in a website, therefore we will exclude patients with no regular access to the Internet or who are unable to fill out forms on the web or navigate websites. We will exclude patients who are unable to walk unassisted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially eligible patients who are planning to initiate chemotherapy for breast cancer will be identified through the Breast Care Clinic. Our power calculation is based on the proportion of patients who successfully complete the study, defined as ≥70% of participants wearing the Fitbit and completing the post-chemotherapy follow-up assessment. Using a 1-sided 1-sample binomial test with α = 0.05, 50 patients, an expected successful completion proportion of 70%, we will have 80% power to reject the null hypothesis if 53% or fewer participants successfully complete the protocol. In other words, the intervention will be considered feasible if 27 or more participants in complete the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence | 9 months
  Adherence, defined at the percentage of weeks that a participant successfully syncs their Fitbit at least once a week during the course of the study, will be reported as a point estimate and 95% confidence interval

SECONDARY OUTCOMES:
Quality of Life - Physical Function | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS physical functioning questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Anxiety | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS anxiety questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Depression | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS depression questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Fatigue | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS fatigue questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Applied cognition general concerns | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS applied cognition general concerns questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Social roles | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS social roles questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Applied cognitive abilities | 12 months from start of chemotherapy
  Mean of PROMIS applied cognitive abilities questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Sleep disturbance | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS sleep disturbance questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Sleep-related impairment | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS sleep-related impairment questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Pain interference | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of PROMIS pain interference questionnaire scores at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported
Quality of Life - Exercise Vital Sign | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Mean of the Exercise Vital Sign (A patient reported measure of the average minutes of moderate or greater physical activity they engage in per week) at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and 6 months following chemotherapy will be reported.
Body Size | Baseline, midpoint of chemotherapy, end of chemotherapy, and 6 months following end of chemotherapy.
  Body mass index (BMI) will be calculated at baseline, midpoint of chemotherapy (This time-point is variable based on drug type, for example, if patient is on a 24 week regimen, midpoint would be distributed at week 12), end of chemotherapy, and at 6 months following chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Melisko, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irwin ML, Crumley D, McTiernan A, Bernstein L, Baumgartner R, Gilliland FD, Kriska A, Ballard-Barbash R. Physical activity levels before and after a diagnosis of breast carcinoma: the Health, Eating, Activity, and Lifestyle (HEAL) study. Cancer. 2003 Apr 1;97(7):1746-57. doi: 10.1002/cncr.11227. PMID 12655532
- [Background] DeSantis CE, Lin CC, Mariotto AB, Siegel RL, Stein KD, Kramer JL, Alteri R, Robbins AS, Jemal A. Cancer treatment and survivorship statistics, 2014. CA Cancer J Clin. 2014 Jul-Aug;64(4):252-71. doi: 10.3322/caac.21235. Epub 2014 Jun 1. PMID 24890451
- [Background] Byar KL, Berger AM, Bakken SL, Cetak MA. Impact of adjuvant breast cancer chemotherapy on fatigue, other symptoms, and quality of life. Oncol Nurs Forum. 2006 Jan 1;33(1):E18-26. doi: 10.1188/06.ONF.E18-E26. PMID 16470230
- [Background] Demark-Wahnefried W, Peterson BL, Winer EP, Marks L, Aziz N, Marcom PK, Blackwell K, Rimer BK. Changes in weight, body composition, and factors influencing energy balance among premenopausal breast cancer patients receiving adjuvant chemotherapy. J Clin Oncol. 2001 May 1;19(9):2381-9. doi: 10.1200/JCO.2001.19.9.2381. PMID 11331316
- [Background] de Jong N, Courtens AM, Abu-Saad HH, Schouten HC. Fatigue in patients with breast cancer receiving adjuvant chemotherapy: a review of the literature. Cancer Nurs. 2002 Aug;25(4):283-97; quiz 298-9. doi: 10.1097/00002820-200208000-00004. PMID 12181497
- [Background] Schwartz AL. Exercise and weight gain in breast cancer patients receiving chemotherapy. Cancer Pract. 2000 Sep-Oct;8(5):231-7. doi: 10.1046/j.1523-5394.2000.85007.x. PMID 11898235
- [Background] Kroenke CH, Chen WY, Rosner B, Holmes MD. Weight, weight gain, and survival after breast cancer diagnosis. J Clin Oncol. 2005 Mar 1;23(7):1370-8. doi: 10.1200/JCO.2005.01.079. Epub 2005 Jan 31. PMID 15684320
- [Background] Schwartz AL, Mori M, Gao R, Nail LM, King ME. Exercise reduces daily fatigue in women with breast cancer receiving chemotherapy. Med Sci Sports Exerc. 2001 May;33(5):718-23. doi: 10.1097/00005768-200105000-00006. PMID 11323538
- [Background] Anderson RT, Kimmick GG, McCoy TP, Hopkins J, Levine E, Miller G, Ribisl P, Mihalko SL. A randomized trial of exercise on well-being and function following breast cancer surgery: the RESTORE trial. J Cancer Surviv. 2012 Jun;6(2):172-81. doi: 10.1007/s11764-011-0208-4. Epub 2011 Dec 10. PMID 22160629
- [Background] Courneya KS, Segal RJ, McKenzie DC, Dong H, Gelmon K, Friedenreich CM, Yasui Y, Reid RD, Crawford JJ, Mackey JR. Effects of exercise during adjuvant chemotherapy on breast cancer outcomes. Med Sci Sports Exerc. 2014 Sep;46(9):1744-51. doi: 10.1249/MSS.0000000000000297. PMID 24633595
- [Background] Ibrahim EM, Al-Homaidh A. Physical activity and survival after breast cancer diagnosis: meta-analysis of published studies. Med Oncol. 2011 Sep;28(3):753-65. doi: 10.1007/s12032-010-9536-x. Epub 2010 Apr 22. PMID 20411366
- [Background] Chasan-Taber S, Rimm EB, Stampfer MJ, Spiegelman D, Colditz GA, Giovannucci E, Ascherio A, Willett WC. Reproducibility and validity of a self-administered physical activity questionnaire for male health professionals. Epidemiology. 1996 Jan;7(1):81-6. doi: 10.1097/00001648-199601000-00014. PMID 8664406